CLINICAL TRIAL: NCT02538939
Title: Efficacy and Tolerance of Sodium Thiosulfate Injection After Ultrasound-guided Percutaneous Irrigation of Calcific Tendinopathy of the Rotator Cuff
Acronym: THIOCAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC14_0394
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Calcific Tendinitis of the Rotator Cuff
Keywords: Calcific tendinitis, Shoulder, Needle lavage, Sodium thiosulfate
MeSH Terms: interventions — sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injection of sodium thiosulfate (Experimental): Needling and lavage of calcific tendinitis of the rotator cuff followed by the injection of sodium thiosulfate
  Interventions: Drug: Sodium thiosulfate

INTERVENTIONS:
Drug: Sodium thiosulfate

SUMMARY:
Calcific tendinitis of the rotator cuff is a common cause of chronic pain of the shoulder. US- guided needling and lavage of the calcification is one of the therapeutic options after failure of conservative management with physiotherapy and anti-inflammatory drugs. The goal of this procedure is to remove the calcific deposit that is believed to cause the sub-acromial impingement. However, studies have shown that complete and rapid disappearance of the calcification deposit after irrigation is rare. The treatment is thought to promote the spontaneous resorption that occurs the weeks and months after the procedure. However, due to this slow process, time to complete recovery can be long. Moreover, it has been shown an association between the amount of removed calcium and improved outcome. Therefore, there is a need to find a way to remove quickly and completely the calcific deposit after irrigation. Sodium thiosulfate has been used successfully in the treatment of calciphylaxis and subcutaneous calcification deposit. The mechanism of action involves chelation of calcium into calcium thiosulfate salts which are much more soluble than other salts of calcium. Our hypothesis is that injection of sodium thiosulfate after irrigation of the calcification will help to dissolve the calcific deposit and thus prompt the disappearance of the calcification.

ELIGIBILITY:
Critères d'inclusion :

* Patients de plus de 18 ans
* Patients affiliés à un régime de sécurité sociale
* Consentement éclairé et signé des patients
* Douleur de l'épaule depuis plus de 3 mois
* Douleur compatible avec une origine péri-articulaire :

  * aggravation lors de l'élévation de l'épaule
  * 1 des 3 tests de conflit sous-acromial positif (Yocum, Hawkins, Neer)
* Présence d'une calcification dure > 5 mm sur la radiographie standard (calcification de type A de la société Française d'Arthroscopie) (Mole, 1993)
* Contraception efficace obligatoire pour les femmes en âge de procréer à maintenir jusqu'au lendemain de l'administration du thiosulfate de sodium.

Critères de non-inclusion :

* Allergie connue à l'anesthésique, au cortivazol ou au thiosulfate de sodium
* Hypersensibilité connue au métabisulfite de sodium (agent de conservation et anti-oxydant connu sous le code E224)
* Patients asthmatiques
* Insuffisance rénale (Clairance < 30 mL/min)
* Patients sous anticoagulants, troubles de la coagulation
* Tableau de résorption aiguë de la calcification (épaule aiguë hyperalgique)
* Aspect flou de la calcification sur les radiographies standards évoquant une résorption (calcification de type C de la société Française d'Arthroscopie) (Mole, 1993) ou calcifications fragmentées à contours nets (type B)
* Rupture de la coiffe des rotateurs mise en évidence sur l'échographie initiale
* Antécédent de PFL sur la calcification étudiée dans les 3 mois précédent l'inclusion
* Autre pathologie d'épaule associée (arthrose gléno-humérale, acromio-claviculaire),
* Diabète déséquilibré
* Contre-indication à la prise d'anti-inflammatoires non stéroïdiens et de paracétamol
* Infection locale ou générale, ou suspicion d'infection
* Contre-indication à la Xylocaïne 1% : (porphyrie récurrente, β-bloquant dans l'insuffisance cardiaque)
* Femmes enceintes, mineurs, majeurs sous tutelle
* Femmes en âge de procréer refusant de maintenir une contraception efficace jusqu'au lendemain de la PFL
* Patients participant à un autre protocole de recherche clinique (à l'exception de recherches non-interventionnelles)
* Patients incapables de suivre le protocole, selon le jugement de l'investigateur

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Decrease the size of the calcific deposit after the PFL | 1 month
  Percentage of patient having more than 50% decrease in the size of the calcific deposit 1 month after the PFL

SECONDARY OUTCOMES:
VAS pain during daily activity (0-10) | 7 days, 1 month and 3 months
VAS pain at rest (0-10) | 7 days, 1 month and 3 months
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | 1 month and 3 months
Size of the calcific deposit assessed by X-Ray of the affected shoulder | 7 days, 1 month and 3 months
Size of the calcific deposit assessed by ultrasound of the affected shoulder | 7 days, 1 month and 3 months
Self-reported quality of life assessed by the EQ-5D questionnaire | 1 month and 3 months
Number of day off work due to the shoulder pain | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

REFERENCES:
- [Derived] Darrieurtort-Laffite C, Bertrand-Vasseur A, Garraud T, Planche L, Le Goff B. Tolerance and effect of sodium thiosulfate in calcific tendinitis of the rotator cuff. Clin Rheumatol. 2020 Feb;39(2):561-569. doi: 10.1007/s10067-019-04793-x. Epub 2019 Nov 1. PMID 31673978